CLINICAL TRIAL: NCT02727595
Title: Evaluation of CyclaPlex Implant for Correction of First Inter Metatarsal Angle in Subjects Suffering From Hallux Valgus Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Cycla Orthopedics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-19-15
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyclaPlex Implant (Experimental): Implant device for reduction of the inter metatarsal angle (IMA) without osteotomy.
  Interventions: Device: CyclaPlex Implant

INTERVENTIONS:
Device: CyclaPlex Implant — Button and suture type implant that will be implanted between the first and second metatarsal

SUMMARY:
The purpose of the study is to evaluate safety, tolerability and performance of the CyclaPlex implant, a button and suture type implant device and instruments for the correction of the first inter metatarsal angle in subjects suffering from Hallux Valgus deformity.

ELIGIBILITY:
Inclusion Criteria:

* Weight less than 100 kilos
* IMA greater than 12 degrees
* IMA less than 7 degrees

Exclusion Criteria:

* Diabetics
* Known osteoporosis
* Known allergy or hypersensitivity to metals
* Gout or any systemic inflammatory arthropathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
IMA Reduction | One year
  The IMA angle is measured pre-op and post-op on x-ray images using internal software. The IMA at end of study should be less than 10 degrees or a reduction of more than 5 degrees.

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) Score | One year
  General improvement as assessed by AOFAS Hallux Scale metatarsophalangeal interphalangeal scale score

CONTACTS AND LOCATIONS:
Overall Officials: Ori Hadash, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No